CLINICAL TRIAL: NCT03750994
Title: Economic Evaluation of Innovative Molecular Analyses in Onco-haematology (PRME-K 2016)
Brief Title: Economic Evaluation of Innovative Molecular Analyses in Onco-haematology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RuBIH2
Record Dates: First submitted 2017-08-11; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Haematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the impact of innovative molecular diagnostics on the clinical management of patients with haematological malignancies via updated Appropriate-Prescribing-Guides including Next-Generation Sequencing (NGS) panels, facilitated therapeutic orientation, and optimised use of costly novel therapeutics and risk-adapted treatment. A micro-costing approach will be used to develop flat fee tarifs for NGS analyses.

DETAILED DESCRIPTION:
The 12 somatic genetic cancer tests that have received temporary authorisation in France form the basis of this study. These tests are not yet in the national biology reimbursement nomenclature but are supported by the ministry of health in a temporary list "Le référentiel des actes innovants hors nomenclature de biologie et d'anatomocytopathologie" (RIHN).

The PRME RuBIH2 will focus on 5 clinical situations in onco-haematology:

1. Myelodysplasia (MDS)
2. Acute lymphocytic leukemia (T) (ALL)
3. Lymphoproliferative disorders (LPD)
4. Acute myeloblastic leukemia (AML)
5. Myeloproliferative disorders (MPD)

The project is organised in 4 complementary work packages (WP): WP1 Cost evaluation, WP2 Prescription Guidelines, WP3 Clinical Validation and WP4 Budget Impact and Organisation.

WP1 will provide costing information on molecular tests and will build on previous studies conducted in France.

WP2 will update existing prescription guidelines based on evidence from the literature and evidence from the WP3. These prescription guidelines will in turn be valued and provide recommendations for a flat fee bundle for pre-specified clinical situations.

WP3 will provide evidence on the clinical impact of molecular diagnosis (in particular NGS) in the 5 pre-specified conditions. Changes in patient management will be measured using a prospective questionnaire for an estimated 3960 molecular tests. The impact of the test on the patient clinical pathway will be analysed. The impact of molecular tests on patient outcome will not be measured.

WP4 will use information from WP1 and WP2 to estimate the budget impact and to provide scenario analyses on the territorial organisation of molecular biology platforms. Based on the estimation of the national activity of molecular onco-haematology platforms the annual functioning budget required to implement molecular diagnosis in France will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematological malignancies referred for molecular diagnosis workup. RuBIH2 will focus on 5 clinical situations in onco-haematology:

  1. Myelodysplasia (MDS)
  2. Acute lymphocytic leukemia (T) (ALL)
  3. Lymphoproliferative disorders (LPD)
  4. Acute myeloblastic leukemia (AML)
  5. Myeloproliferative disorders (MPD)

Exclusion Criteria:

* Other haematological diseases not included in the list above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for molecular diagnosis at one of the certified molecular onco-haematology platforms in France.
Sampling Method: Non-Probability Sample
Enrollment: 3960 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Next Generation Sequencing (NGS) tests that have a clinical impact for the patient for five hematological malignancies. | 2 years
Percentage of Next Generation Sequencing (NGS) that are from the oncologists internal to the platform versus external centres. | 2 years
Average time in days between the Next Generation Sequencing (NGS) prescription being issued and the results being rendered to the clinician. | 2 years
Percentage of prescriptions for diagnostics, prognostic, theranostics or treatment response | 2 years
Percentage of the genetic targets that are analysed for research purposes versus immediate clinical utility for the patient. | 2 years
Percentage of patients prescribed the Next Generation Sequencing (NGS) at the diagnostic stage or before second (or higher) line treatment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Claude Preudhomme, Professor, Principal Investigator — DRCI AP-HP
Locations (26):
- France (26):
  - Centre hospitalier régional universitaire de Lille, Lille, Hauts-de-France
  - CHU Angers, Angers
  - Hôpital Avicenne AP-HP, Bobigny
  - CHU de Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Henri Mondor AP-HP, Créteil
  - CHRU Dijon Bourgogne, Dijon
  - CHU Limoges, Limoges
  - CHU Lyon Sud Pierre Bénite, Lyon
  - CHU Montpellier, Montpellier
  - CHU Hôtel Dieu, Nantes
  - CHU Nice, Nice
  - Hôpital Pitié-Salpêtrière AP-HP, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital St Louis AP-HP, Paris
  - Hôpital Cochin AP-HP, Paris
  - Hôpital Necker AP-HP, Paris
  - Hôpital Saint Antoine AP-HP, Paris
  - CHU Robert Debré Reims, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri-Becquerel, Rouen
  - Centre hospitalier universitaire de Saint-Étienne, Saint-Etienne
  - Hôpitaux Universitaires Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - Institut Gustave Roussy, Villejuif